CLINICAL TRIAL: NCT04040855
Title: The Impact of Medication Reviews Conducted in Primary Care on Hospital Admissions and Mortality - a Randomized Controlled Trial
Brief Title: Medication Reviews in Elderly in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2018/8
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Drug Utilization Review
Keywords: medication reviews, elderly, primary care
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Patients were blindly randomized to intervention or control group in 2011. This study is a follow-up with additional data collection for the included patient, a total of 369.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Closed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention groups received multi-professional medication reviews. A nurse performed a symptom evaluation, a pharmacist assessed the drug list and made adjustment suggestions and finally a physician took action and performed medication changes.
  Interventions: Other: Medication review
- Control (No Intervention): Patients were treated according to the usual routine.

INTERVENTIONS:
Other: Medication review — Multi-professional medication review
  Arms: Intervention

SUMMARY:
The study is a follow-up of a randomized controlled study performed in 2011-2012 with medication reviews in elderly patients in Sweden. Additional data about mortality and hospital admissions have been collected.

DETAILED DESCRIPTION:
Background Drug-related problems among the elderly population are common and increasing. Multi-professional medication reviews (MR) have arisen as a method to optimize drug therapy for frail elderly patients. Research has not yet been able to show conclusive evidence of the effect of MRs on mortality or hospital admissions. Aim The aim of this study was to assess the impact of MRs' on hospital admissions and mortality after six and 12 months in a frail population of 369 patients in primary care in a randomized controlled study. Methods Patients were blindly randomized to an intervention group (receiving MRs) and a control group (receiving usual care). Descriptive data on mortality and hospital admissions at six and 12 months were collected. Survival analysis was performed for time to death and time to the first hospital admission within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* age>75 years, living in nursing homes or community-dwelling with municipality-provided care, with multi-dose drug dispensing

Exclusion Criteria:

* lack of multi-dose drug dispensing, living at home with no municipality-provided care, <75 years old

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 369 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
hospital admission | six months
  time to the first hospital admission
hospital admission | twelve months
  time to the first hospital admission
Survival analysis | six months
  time to death
Survival analysis | twelve months
  time to death

SECONDARY OUTCOMES:
number of hospital admissions | six months
  number of hospital admissions
number of hospital admissions | twelve months
  number of hospital admissions
mortality | six months
  number of deaths
mortality | twelve months
  number of deaths

OTHER OUTCOMES:
number of drugs | base-line
  number of drugs

REFERENCES:
- [Derived] Milos Nymberg V, Lenander C, Borgstrom Bolmsjo B. The Impact of Medication Reviews Conducted in Primary Care on Hospital Admissions and Mortality: An Observational Follow-Up of a Randomized Controlled Trial. Drug Healthc Patient Saf. 2021 Jan 27;13:1-9. doi: 10.2147/DHPS.S283708. eCollection 2021. PMID 33536791